CLINICAL TRIAL: NCT00387400
Title: A Phase I Study of Temozolomide and RAD001C in Patients With Malignant Glioblastoma Multiforme
Brief Title: Temozolomide + Everolimus in Newly Diagnosed, Recurrent, or Progressive Malignant Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I162; CAN-NCIC-IND162 (Registry Identifier: PDQ); CDR0000507616 (Other: PDQ)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult gliosarcoma; recurrent adult brain tumor; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Everolimus; Temozolomide; Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: everolimus — 150 mg/m2/day PO Daily x 5, q 4 weeks
Drug: temozolomide — 2.5 mg PO Daily, beginning day 2 of cycle 1, q 4 weeks
Genetic: microarray analysis — Tissue sections will be stained by immunohisto-chemistry using the following antibodies: EGFRvIII, PTEN, phospho-specific PKB/Akt Ser473; phosphor-mTORSer2448, p70S6K Thr389; S6 ribosomal protein Ser235/236. These antibodies are selected on the basis of providing a readout of upstream and downstream signaling through mTOR, and availability of antibodies that reliably stain paraffinembedded tissue.
Other: immunohistochemistry staining method — Tissue sections will be stained by immunohisto-chemistry using the following antibodies: EGFRvIII, PTEN, phospho-specific PKB/Akt Ser473; phosphor-mTORSer2448, p70S6K Thr389; S6 ribosomal protein Ser235/236. These antibodies are selected on the basis of providing a readout of upstream and downstream signaling through mTOR, and availability of antibodies that reliably stain paraffinembedded tissue.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving temozolomide together with everolimus may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of everolimus when given together with temozolomide in treating patients with newly diagnosed, recurrent, or progressive malignant glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose(s) and the recommended phase II dose(s) of everolimus when administered with standard-dose temozolomide in patients with newly diagnosed, recurrent, or progressive glioblastoma multiforme.
* Determine the toxicity of this regimen in these patients.

Secondary

* Determine the efficacy of this regimen in patients with measurable disease at baseline.
* Identify correlates of activity by molecular study of paraffin-embedded tumor samples from these patients.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a nonrandomized, nonblinded, parallel-group, multicenter, dose-escalation study of everolimus. Patients are stratified according to concurrent use of enzyme-inducing antiepileptic drugs (yes vs no).

Patients receive oral temozolomide once daily on days 2-5 in course 1 and on days 1-5 in all subsequent courses. Patients also receive oral everolimus once daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients with newly diagnosed disease receive up to 6 courses of treatment. Patients with recurrent disease who achieve a response (partial or complete response) or stable disease may continue treatment until disease progression or unacceptable toxicity.

Cohorts of 3-6 patients per stratum receive escalating doses of everolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during the first course of therapy. Once the MTD is determined, an additional 6 patients are treated at the MTD.

Patients' archival diagnostic tumor tissue is evaluated during study for correlative molecular studies (by immunohistochemical staining) of mammalian target of rapamycin inhibition status (mTOR activity) and pretreatment molecular markers. Blood samples are taken periodically during course 1 for pharmacokinetic studies.

After completion of study therapy, patients are followed at 4 weeks. Patients with stable or responding disease are then followed every 3 months until relapse or progression.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioblastoma multiforme, meeting 1 of the following criteria:

  * Newly diagnosed disease AND meets the following criteria:

    * Has undergone prior surgery and radiotherapy with concurrent temozolomide
    * No prior chemotherapy except for concurrent low-dose temozolomide given with radiotherapy
  * Recurrent or progressive disease after front-line therapy AND meets the following criteria:

    * No more than 1 prior chemotherapy regimen in the adjuvant setting
    * More than 4 months since last adjuvant treatment
    * No prior chemotherapy for recurrence
* Bidimensionally measurable disease, defined as ≥ 1 enhancing lesion ≥ 1 cm x 1 cm by CT scan or MRI, within 21 days of study entry (for patients with recurrent/relapsed disease)

  * Patients receiving steroids must be on stable dose for at least 14 days before baseline CT scan or MRI
* Paraffin-embedded sample of primary or metastatic tumor diagnostic specimen must be available

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 120,000/mm³
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No upper gastrointestinal condition or other condition that would preclude compliance with oral medication
* No other prior malignancy except for adequately treated nonmelanoma skin cancer, curatively treated in situ cervical cancer, or other solid tumors curatively treated with no evidence of disease for the past 5 years
* No serious illness or underlying medical condition that would preclude study compliance, including any of the following:

  * Significant neurologic or psychiatric disorder that would preclude obtaining informed consent
  * Active, ongoing infection
* No known hypersensitivity to everolimus or temozolomide or their components

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 weeks since prior surgery and recovered
* At least 4 weeks since prior radiotherapy
* Concurrent enzyme-inducing antiepileptic drugs allowed
* No concurrent inhibitors of cytochrome 3A4 (e.g., ketoconazole and similar antifungals, erythromycin, or diltiazem)
* No other concurrent experimental drugs, anticancer treatment, or investigational therapy
* No concurrent grapefruit juice

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-03-20 (Actual); Primary Completion 2010-09-24 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of everolimus as measured by NCI CTCAE v3.0 | from the time of the first treatment

SECONDARY OUTCOMES:
Response as measured by CT scan and/or brain MRI at baseline and after every other course and clinical neurologic assessment at baseline and after every course | after every other course
Correlation of clinical outcome with pretreatment tumor tissue molecular markers as measured by molecular studies of paraffin-embedded tumor samples | 4 years
  Assessed at study completion
Pharmacokinetics of everolimus during course 1 | during course 1

CONTACTS AND LOCATIONS:
Overall Officials: Warren P. Mason, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (9):
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mason WP, Macneil M, Kavan P, Easaw J, Macdonald D, Thiessen B, Urva S, Lwin Z, McIntosh L, Eisenhauer E. A phase I study of temozolomide and everolimus (RAD001) in patients with newly diagnosed and progressive glioblastoma either receiving or not receiving enzyme-inducing anticonvulsants: an NCIC CTG study. Invest New Drugs. 2012 Dec;30(6):2344-51. doi: 10.1007/s10637-011-9775-5. Epub 2011 Dec 9. PMID 22160854